CLINICAL TRIAL: NCT03650309
Title: Deep Brain Stimulation for the Treatment of Refractory Morbid Obesity
Brief Title: Deep Brain Stimulation for Morbid Obesity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Principal Investigator, Andres M. Lozano, Neurosurgeon, Professor of Surgery, University Health Network, Toronto
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 17-5899
Record Dates: First submitted 2018-08-10; First posted 2018-08-28 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Obesity; Obesity, Morbid
Keywords: Deep Brain Stimulation; Functional Neurosurgery; Neuromodulation; Bariatrics; Weight Loss; Addiction
MeSH Terms: conditions — Obesity; Obesity, Morbid; Weight Loss; Behavior, Addictive | interventions — Deep Brain Stimulation

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Deep Brain Stimulation (Experimental): All patients will receive deep brain stimulation (DBS) targeting two brain areas involved in the pathophysiology of obesity. No other changes to pre-existing treatment will be made. This is the only arm in this experiment.
  Interventions: Device: Deep Brain Stimulation

INTERVENTIONS:
Device: Deep Brain Stimulation — All patients will undergo surgical implantation of a deep brain stimulation (DBS) system, which involves placement of stimulating electrodes in the brain. These electrodes will be used to deliver electrical current to target two brain structures involved in the pathophysiology of obesity.

SUMMARY:
This is an open-label, phase I pilot trial designed to evaluate the safety and feasibility of deep brain stimulation (DBS) for the treatment of refractory morbid obesity. Patients with diagnoses of morbid obesity will be recruited and enrolled. All patients will receive DBS targeting two brains areas involved in the pathophysiology of obesity and will be followed post-operatively for 12 months.

DETAILED DESCRIPTION:
This study will establish 1)the safety of deep brain stimulation (DBS) in a patient population with treatment refractory morbid obesity. DBS has been used safely and effectively in thousands of patients for numerous disorders. Recent evidence (outlined above) has shown that DBS can also be used to manage refractory psychiatric conditions, such as depression and obsessive-compulsive disorder, as well as in eating disorders such as anorexia nervosa. Such studies indicate that a targeted therapy informed by the neuroanatomic and circuitry literature can be effective in altering pathological mood and behaviour. 2) evaluate the effectiveness of the procedure, which will be evaluated by the actual weight loss and resolution of the core symptoms of morbid obesity, including BMI, as well of, depression, self-esteem, and binge eating scores surrounding with loss or weight gain.

ELIGIBILITY:
Inclusion Criteria:

1. Female or Male patients between age 20-60
2. Diagnosis of Morbid Obesity (defined as a BMI>40kg/m2 or BMI>35 with 1 obesity related comorbidity) OR a diagnosis of Binge Eating Disorder not responsive to recommended treatments (as defined by the DSM-5)
3. Failure or non eligibility of bariatric surgery with <50% of excess weight loss, with or without BMI>35 kg/m2, at 18 months or more after the operation; OR diagnosis of binge eating disorder for over 18 months
4. Diagnosis of food dependence via Yale Food Addiction Scale (YFAS) criteria
5. Normal neurological exam
6. Normal head CT scan and cerebral MRI
7. Patient informed and able to give written consent
8. Able to comply with all testing, follow-ups and study appointments and protocols

Exclusion Criteria:

1. Active neurologic disease such as epilepsy
2. Alcohol or substance dependence or abuse in the last 6 months, excluding caffeine and nicotine
3. Any contraindication to magnetic resonance imaging (MRI) or positron emission tomography (PET) scanning
4. Likely to relocate or move during the study's one year duration
5. Presence of cardiac arrhythmias, or other cardiac, respiratory, renal or endocrine conditions as a result of morbid obesity, that will result in significant risk from a surgical procedure.
6. Presence of epilepsy, stroke or degenerative disorder of the nervous system
7. Pregnancy

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2018-09-01 (Actual); Primary Completion 2022-01-23 (Actual); Study Completion 2022-07-23 (Actual)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events | 12 months
  Patients will be closely monitored for adverse events following DBS surgery with regular check-ups.

SECONDARY OUTCOMES:
Weight | 12 months
  Weight (in kilograms) will be frequently assessed prior to and following DBS surgery.
'Quality of Life Scale' Questionnaire | 12 months
  Patients will regularly complete the 16-item Quality of Life Scale questionnaire (worst score = 16, best score = 112) to assess psychosocial function.
'Behavioral Inhibition System/Behavioral Activation System Scales (BIS/BAS Scales)' Questionnaire | 12 months
  Patients will regularly complete the 24-item BIS/BAS Scales questionnaire to assess psychosocial behaviour. This questionnaire has 3 sub-scales: 'BAS drive' (highest score = 16, lowest score = 4), 'BAS fun seeking' (highest score = 20, lowest score = 5), 'BAS reward responsiveness' (highest score = 20, lowest score = 5), and 'BIS' (highest score = 28, lowest score = 7).
'Patient Health Questionnaire (PHQ-9)' Questionnaire | 12 months
  Patients will regularly complete the 9-item PHQ-9 questionnaire (worst score = 27, best score = 0) to assess mood and depression symptoms.
'Generalized Anxiety Disorder 7-item (GAD-7)' Questionnaire | 12 months
  Patients will regularly complete the 7-item GAD-7 questionnaire (worst score = 21, best score = 0) to assess anxiety symptoms.
'Difficulties in Emotion Regulation Scale (DERS)' Questionnaire | 12 months
  Patients will regularly complete the 36-item DERS questionnaire (worst score = 180, best score = 36) to assess emotional dysregulation.
'Yale-Brown Obsessive Compulsive Scale (Y-BOCS)' Questionnaire | 12 months
  Patients will regularly complete the 10-item Y-BOCS questionnaire (worst score = 40, best score = 0) to assess severity of obsessive and compulsive symptoms
'Binge Eating Scale (BES)' Questionnaire | 12 months
  Patients will regularly complete the 16-item BES questionnaire (worst score = 43, best score = 0) to assess binge eating symptoms
'Yale-Brown-Cornell Eating Disorder Scale (YBC-EDS)' Questionnaire | 12 months
  Patients will regularly complete the 19-item YBC-EDS questionnaire (worst score = 32, best score = 0) to assess eating-related preoccupations and rituals
'Emotional Eating Scale (EES)' Questionnaire | 12 months
  Patients will regularly complete the 25-item EES questionnaire (worst score = 100, best score = 0) to assess their emotional relationship with food.
'Power of Food (POF)' Questionnaire | 12 months
  Patients will regularly complete the 15-item POF questionnaire (worst score = 75, best score = 15) to assess the degree of influence food exerts on their day-to-day life.
'Eating Disorder Examination Questionnaire (EDE-Q)' | 12 months
  Patients will regularly complete the 28-item EDE-Q (worst score = 6, best score = 0) to assess aspects of eating behaviour including restraint, eating concern, shape concern, and weight concern.
'Yale Food Addiction Scale (YFAS)' Questionnaire | 12 months
  Patients will regularly complete the 25-item YFAS (higher numbers = more severe symptoms) to assess the severity of food addiction.

CONTACTS AND LOCATIONS:
Overall Officials: Andres Lozano, Principal Investigator — University Health Network, Toronto
Locations (1):
- Toronto Western Hospital, University Health Network, Toronto, Ontario, Canada